CLINICAL TRIAL: NCT05599698
Title: Effects of Chemotherapy on Perceived Daily Performance and Executive Functions of Adults With Cancer
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bnai Zion Medical Center (Other Government)
Collaborators: Tel Aviv University (Other)
Responsible Party: Principal Investigator, abed.agbarya, Dr., Bnai Zion Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0106-22-BNZ
Record Dates: First submitted 2022-10-26; First posted 2022-10-31 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cancer
Keywords: executive functioning; daily functioning; chemotherapy; non-central nervous system malignancy
MeSH Terms: conditions — Neoplasms | interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- chemotherapy (Experimental): chemotherapy
  Interventions: Other: Chemotherapy

INTERVENTIONS:
Other: Chemotherapy — Standard chemotherapy protocols for adjuvant & neoadjuvant treatment for different types of solid malignancies

SUMMARY:
The purpose of this study is to examine changes in perceived daily performance and executive functioning following chemotherapy in individuals with non-central nervous system cancers.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed with a primary non-central nervous system malignancy (lung, breast, colon, ulcer, urinary tract, canine tumors).
* Stages I-III.
* Pre-commencement of adjuvant (post-surgery) or neoadjuvant (prior to surgery) chemotherapy.
* Understand and read Hebrew.
* Have at least 12 years of education.

Exclusion Criteria:

* Diagnosed with central nervous system malignancies.
* Had a previous malignancy.
* Have or had metastatic disease.
* Have a history of a neurological condition or severe depression.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-11-15 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in scores of Canadian Occupational Performance Measure. | Change between Pre-to post (three months) chemotherapy
  Canadian Occupational Performance Measure - COPM assesses perceived daily performance and performance satisfaction with meaningful daily activities.
  During the pre-chemotherapy assessment, participants will identify up to five activities that they prioritize as meaningful for them. Each of these activities is then rated on a 10-point scale for perceived performance (1=not able to do at all, 10=able to do extremely well) and similarly for satisfaction with performance. The final scores of the COPM are the average scores for total performance and for satisfaction (higher scores indicate better performance or satisfaction with performance). During the post-chemotherapy assessment, the participants will rate the same activities they prioritized in the pre-chemotherapy assessment.

SECONDARY OUTCOMES:
Reintegration to Normal Living index. | Change between Pre-to post (three months) chemotherapy
  Assesses daily participation in recreational and social activities, movement within the community, and degree of comfort the individual has in his/her role in the family and with other relationships.
Backward Digit Span. | Change between Pre-to post (three months) chemotherapy
  Assesses working memory capacity
Dual Tasking by performing two tasks concurrently (motor by the Box & Blocks Test and cognitive by backward subtraction for one minute) | Change between Pre-to post (three months) chemotherapy
  Assesses dual tasking by performing two tasks concurrently
Color Trail Test - CTT | Change between Pre-to post (three months) chemotherapy
  Assesses cognitive flexibility
Cognitive performance-based assessment will be assessed by the Weekly Calendar Planning Activity. | Change between Pre-to post (three months) chemotherapy
  A performance-based assessment that examines the influence of subtle executive function difficulties on person's ability to perform a multiple-step activity.
Cognitive Self Efficacy FACT-Cognitive Function questionnaire | Change between Pre-to post (three months) chemotherapy
  FACT-Cognitive Function questionnaire Version 3 assesses cognitive functioning in individuals with cancer. For assessing cognitive self-efficacy we will use the cognitive self-abilities subscale (CogPCA) of the questionnaire, which includes 7 statements with responses given on a 5-point Likert scale (from 0, never; to 4, several times a day). The score range= 0-28 with higher scores indicating higher difficulties.
Emotional Well-Being FACT-G questionnaire | Change between Pre-to post (three months) chemotherapy
  Emotional Well-Being will be assessed by the emotional well-being subscale from the FACT-G (General) questionnaire (https://www.facit.org/). The EWB scale includes six statements with responses given on a 5-point Likert scale (from 0, not at all; to 4, very much). The score range= 0-24 with higher scores indicating higher emotional deficits.
Functional Assessment of Chronic Illness Therapy - Fatigue (FACIT-F) | Change between Pre-to post (three months) chemotherapy
  Fatigue will be assessed by the FACIT Fatigue questionnaire FACIT-F, Version 4 which includes 13 statements with responses given on a 5-point Likert scale (from 0, not at all; to 4, very much). The score range= 0-52 with higher scores indicating more fatigue.
Qualitative open-ended questions regarding perceived changes in participants' cognitive functioning following cancer diagnosis and how these changes affect their daily functioning | Pre chemotherapy
  Open ended questions will be presented on a sheet of paper and the participants will be asked to write their answers bellow together with the accessor. Reporting does not include a score on a scale.
Qualitative open-ended questions regarding perceived changes in participants' cognitive functioning following chemotherapy and how these changes affect their daily functioning | Post (three months) chemotherapy
  Open ended questions will be presented on a sheet of paper and the participants will be asked to write their answers bellow together with the accessor. Reporting does not include a score on a scale.

OTHER OUTCOMES:
Demographic and medical data Questionnaire | pre-chemotherapy
  The questionnaire will include the following details: age (years), education (years), sex (female, male), marital status (married, not married, divorced, widow), number of children, work status (employed, not employed, independent), dominant hand (right, left), socioeconomic level (income level), type/stage of cancer (1,2,3), disease characteristics (e.g., size of the tumor, number of affected lymph nodes), details of treatments received (e.g., types of surgery chemotherapy regimens, date of chemo commencement, number of cycles completed).

CONTACTS AND LOCATIONS:
Overall Officials: Abed Agbarya, MD, Principal Investigator — abed.agbarya@b-zion.org.il
Locations (1):
- Bnai Zion Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Articles are planned for publication of the study protocol and final study results.
Supporting Information: Study Protocol, CSR
Time Frame: 24 - 30 months